CLINICAL TRIAL: NCT03873129
Title: Optimizing HIV Care for Patients With Substance Use Disorders Using Predictive Analytics in a Mobile Health Application
Brief Title: ART-CHESS: A Mobile Health Application to Support People Living With HIV and Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1190; A534265 (Other: UW Madison); SMPH\MEDICINE\INFECT DIS (Other: UW Madison); 1DP2DA042424-01 (NIH); Protocol Version 3/20/20 (Other: UW Madison)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2020-06

CONDITIONS: HIV/AIDS; Substance Use Disorders
Keywords: antiretroviral therapy; HIV transmission
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Phase 2 is single group trial of A-CHESS when implemented in 2 high-volume HIV clinics, providing evidence describing the effectiveness and durability of an mHealth strategy for maintaining viral suppression among patients with substance use disorders treated with ART.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A-CHESS (Experimental): participant will be using the A-CHESS mobile app for 12 months
  Interventions: Behavioral: mobile health app (mHealth)

INTERVENTIONS:
Behavioral: mobile health app (mHealth) — A-CHESS is a mobile health app for participants to interact with their treatment team for 12 months.
  Other Names: ART-CHESS

SUMMARY:
It is now well-accepted that lowering community-level viral load through expansion of antiretroviral therapy (ART) can reduce HIV transmission among people who use drugs. However, achieving durable viral suppression among patients with substance use disorders is a major challenge for providers and health systems. This study aims to adapt and implement an existing mobile health (mHealth) system, A-CHESS (Addiction Comprehensive Health Enhancement Support System) to improve care for HIV patients with substance use disorders.

DETAILED DESCRIPTION:
Patients with substance use disorders are continuously at risk for relapse and other disruptive life events, which may lead to lapses in antiretroviral treatment and subsequent viral rebound, thereby increasing their level of infectivity. Behaviors that place others at risk for HIV transmission such as sharing drug paraphernalia and unprotected sex may also increase during these periods of social and behavioral instability.

Various biomedical, behavioral, and structural interventions have been used to prevent lapses in HIV care or minimize their impact when they occur. A potentially transformative strategy would be the one that makes novel use of ubiquitous technology and the existing clinical workforce to provide highly-effective, tailored support to the patients at greatest risk, at the time and place it is needed the most.

This study has 2 phases:

Phase I has been completed and it was an observational study, not a clinical trial. Patients who volunteered were recruited to use the mobile phone app to enter data, but it was not intended to improve their health or health care. The data collected during phase 1 will be used to inform the intervention in phase 2, where the study team hope to use the system to improve patient care.

Phase 2 will conduct a single-arm implementation study (with historical controls) of A-CHESS when implemented in 2 high-volume HIV clinics, providing evidence describing the effectiveness and durability of an mHealth strategy for maintaining viral suppression among patients with substance use disorders treated with ART.

The long-term goal of this project is to develop a comprehensive mHealth system that identifies the critical time-varying determinants of lapses in HIV care for substance using patients, and translates these diverse inputs into actionable, patient-specific alerts to clinical providers. This goal will be achieved by adapting and implementing an existing mHealth intervention, A-CHESS, which might improve HIV care for patients with substance use disorders through two mechanisms. First, existing A-CHESS services will improve treatment adherence by enhancing self-determination (i.e., intrinsic motivation, competence and social relatedness). Second, through new functionality incorporating predictive analytics with patient-level data, A-CHESS will identify moments when patients are at the highest risk for antiretroviral treatment failure, allowing clinic-based staff to provide targeted interventions that maximize the efficiency of care coordination resources.

If successful, this project would translate important individual and neighborhood-level data into timely and clinically-relevant knowledge that is accessible to the HIV care team, representing a major step forward in our ability to support patients with complex needs.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years old
2. Documentation of HIV infection
3. Able to read and write in English
4. A history of substance use disorder, defined as one or more of the following:

   1. A positive result on one or more SUD screening tests (see "Screening," below), reflecting substance use during the prior year.
   2. Current participation in a substance abuse treatment program, including medication assisted treatment for SUD, or regular (at least monthly) participation in SUD-oriented support groups.
   3. A lifetime history of problematic drug or alcohol use AND having been incarcerated in the past year, regardless of the date of last substance use.

Exclusion Criteria:

1. Individuals who are under 18, are not HIV-positive, who have no history of alcohol or drug misuse, or cannot read and write in English
2. Individuals who are prohibited from using the internet on any device as a condition of criminal justice supervision
3. Individuals who cannot demonstrate competency in using the A-CHESS interface on a smartphone or web browser after a standard period of training by a research staff member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Change in the Viral suppression among study semesters of A-CHESS use versus semesters of without A-CHESS use. | Up to 12 months
  Viral suppression will be measured each 6 months period. HIV RNA< 200 copies/mL reflects viral suppression per protocol.

SECONDARY OUTCOMES:
Change in the Attendance at HIV Clinic Appointments among study semesters of A-CHESS use versus semesters of without A-CHESS use. | up to 12 months
  Attendance at HIV clinic appointments
Change in the Drug usage among study semesters of A-CHESS use versus semesters of without A-CHESS use. | up to 12 months
  Change in the Drug usage among study semesters of A-CHESS use versus semesters of without A-CHESS use.
Change in the Medication adherence among study semesters of A-CHESS use versus semesters of without A-CHESS use. | up to 12 months
  Change in the Medication adherence among study semesters of A-CHESS use versus semesters of without A-CHESS use.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Westergaard, MD, PhD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States